CLINICAL TRIAL: NCT01111292
Title: Myo-Inositol Chemoprevention in Colitis-Associated Dysplasia
Brief Title: Inositol in Preventing Colorectal Cancer in Patients With Colitis-Associated Dysplasia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was closed prematurely due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2011-01434; NCI-2011-01434 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000671302; NCI09-13-02 (Other: Northwestern University); NWU09-13-02 (Other: DCP); P30CA060553 (NIH); N01CN35157 (NIH)
Record Dates: First submitted 2010-04-24; First posted 2010-04-27 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Colon Carcinoma; Dysplasia in Crohn Disease; Low Grade Dysplasia in Ulcerative Colitis; Rectal Carcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (inositol) (Experimental): Beginning within 14 days after colonoscopy, patients receive inositol PO QD on days 1-14 and BID on days 15-90.
  Interventions: Drug: Inositol
- Arm II (placebo) (Placebo Comparator): Beginning within 14 days after colonoscopy, patients receive placebo PO QD on days 1-14 and BID on days 15-90.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Inositol — Given PO
  Other Names: myo-Inositol
  Arms: Arm I (inositol)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This pilot, randomized phase I/II trial studies how well inositol works in preventing colorectal cancer in patients with abnormal cells (dysplasia) associated with inflammation of the colon (colitis). Patients with colitis-associated dysplasia may have an increased risk of developing colorectal cancer. Inositol is a vitamin-like substance that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of myo-inositol (inositol), administered for 3 months, on phospho (P)-beta (B)-catenin staining in areas of low-grade dysplasia or in areas of prior low grade dysplasia in subjects with known colitis-induced low grade dysplasia at baseline.

SECONDARY OBJECTIVES:

I. To examine the effect of myo-inositol on regression of dysplasia. II. To examine the effect of inositol on p53 and Ki67 staining within remaining dysplasia.

III. To examine the effect of inositol on epithelial apoptosis (cleaved caspase-3) within dysplasia.

IV. To examine the effect of inositol on reductions in mucosal messenger ribonucleic acid (mRNA) levels of monocyte chemotactic protein 1 (MCP1), inducible nitric oxide synthase (iNOS), and cyclooxygenase (Cox)-2.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Beginning within 14 days after colonoscopy, patients receive inositol orally (PO) once daily (QD) on days 1-14 and twice daily (BID) on days 15-90.

ARM II: Beginning within 14 days after colonoscopy, patients receive placebo PO QD on days 1-14 and BID on days 15-90.

After completion of treatment, patients undergo biopsy and colonoscopy with or without mucosal resection.

After completion of study treatment, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have ulcerative colitis or Crohn's disease with low grade dysplasia or polyploid dysplasia or have a history of dysplasia and increased positive beta-catenin levels confirmed by a consensus of the study pathologists (2 of 2, or 2 of 3)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) > 1,500/uL
* Platelets > 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT] =< 1.5 times upper limit of normal
* Creatinine within normal institutional limits
* International normalized ratio (INR) < 1.5
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of baseline pregnancy test, throughout the duration of the study, and for 1 month following cessation of study drug; females must begin adequate contraception immediately following screening pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; if she is pregnant, she will be immediately withdrawn from the study and followed until the birth of the child
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with life-threatening medical conditions that would preclude study treatment intervention and colonoscopy
* Participants may not be receiving any other investigational agents
* History of allergic reactions to rice or compounds of similar chemical or biologic composition to myo-inositol (i.e., urticaria, dermatologic reaction)
* Use of medications known to elevate serum blood glucose; participants on steroids are still eligible, as they will be monitored weekly for fasting blood glucose
* Participants with dysplasia-associated lesion or mass (DALM), high-grade dysplasia or invasive colonic carcinoma are excluded
* Uncontrolled intercurrent illness including, but not limited to

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Chronic renal failure
  * Chronic renal insufficiency
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Prior treatment with myo-inositol
* History of systemic chemotherapy within 18 months of screening
* Subjects taking valproic acid and/or lithium
* Diabetes mellitus
* History of total proctocolectomy
* Concomitant primary sclerosing cholangitis (PSC)
* Pregnant or lactating subjects are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mount Sinai Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 73 patients were screened for study eligibility. Of those, 68 patients were ineligible (no biopsies were taken from 5 patients and 63 did not have a diagnosis of dysplasia at the initial visit).
Pre-assignment Details: Serum myo-inositol levels were measured from 13 patients who were screened for study eligibility, and those levels (23.28+/-6.46 μM) were consistent with previously published data (Chiu et al, Dolhofer et al, Lewin et al).
Groups:
- Arm I (Inositol): Beginning within 14 days after colonoscopy, patients receive inositol PO QD on days 1-14 and BID on days 15-90.
  Inositol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Placebo): Beginning within 14 days after colonoscopy, patients receive placebo PO QD on days 1-14 and BID on days 15-90.
  Placebo: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Randomization
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Treatment
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Started | 3 | 2
Completed | 2 | 1
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1
Period: Post Treatment Biopsy
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Follow-Up
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Inositol) | Arm II (Placebo) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Myo-inositol (Inositol) on P-β-catenin Staining in Areas of Low Grade Dysplasia in Subjects With Known Colitis-induced Low Grade Dysplasia.
Description: The primary objective of this study will be to evaluate the effect of myo-inositol (inositol), administered for three months, on P-β-catenin staining in areas of low grade dysplasia or in areas of prior low grade dysplasia in subjects with known colitis-induced low grade dysplasia at baseline.
Time Frame: Baseline to 90 days
Population: pβ-cat-positive cell counts in pre- and post-study biopsies with dysplasia or adenoma. Counts are broken down as the number of crypts with 3, 4, or 5 pβ-cat positive cells. High frequency (HF) fields of view are those containing at least 2 crypts with three or more pβ-cat positive cells per crypt (at 20X). I
Measure: Mean (Standard Deviation); unit: Colonic Biopsies
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Number analyzed (Participants) | 2 | 1
Colonic Biopsies
  Baseline Cells/100 IEC | 2.5 (2.5) | 0 (0)
  Post Intervention Cells/100 IEC | 3.67 (.94) | 0
  Baseline Crypts w/2 cells | 7.75 (7.85) | 2.5 (5)
  Post Intervention Crypts w/ 2 cells | 8.67 (2.49) | 0 (0)
  Baseline Crypts w/3 cells | 2 (1.58) | .5 (.5)
  Post Intervention Crypts w/ 3 Cells | 2.67 (1.25) | 0 (0)
  Baseline Crypts w/4 cells | 2 (1.58) | 0 (0)
  Post Intervention Crypts w/4 cells | 1.67 (1.7) | 0 (0)
  Baseline Crypts w/>5 cells | 2.25 (2.28) | 0 (0)
  Post Intervention Crypts w/>5 cells | 0 (0) | 0 (0)
  Baseline # HF Fields of View | 2.5 (2.3) | 0 (0)
  Post Intervention # HF Fields | 2 (.82) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Arm I (Inositol) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Inositol) (N=3) | Arm II (Placebo) (N=2)
Gastrointestinal disorder: Stomach Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal Disorder: Diarrhea (Gastrointestinal disorders) | 1 (20) | 1 (3)
Gastrointestinal disorder: Amal Henorrhage: Blood in sttol (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder: Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder: Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disprder: Hemorroids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Disorder: High Bilirubin (Investigations) | 1 (1) | 0 (0) — Blood bilirubin increased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less